CLINICAL TRIAL: NCT07094009
Title: Comparison of the Clinical Efficacy and Adverse Reactions of Different Needling Patterns of High-frequency Microneedles in the Treatment of Axillary Odor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Chengcheng Shen, Attending Physician of Dermatology, First Affiliated Hospital of Chongqing Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-435
Record Dates: First submitted 2025-07-23; First posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Axillary Hyperhidrosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- transverse needling group (Experimental): received transverse needling
  Interventions: Procedure: received transverse needling
- vertical needling group (Experimental): received vertical needling
  Interventions: Procedure: received vertical needling
- mixed needling group (Experimental): received mixed needling
  Interventions: Procedure: received mixed needling

INTERVENTIONS:
Procedure: received transverse needling — received transverse needling of high-frequency microneedles
  Arms: transverse needling group
Procedure: received vertical needling — received vertical needling of high-frequency microneedles
  Arms: vertical needling group
Procedure: received mixed needling — received mixed needling of high-frequency microneedles
  Arms: mixed needling group

SUMMARY:
* Background: Axillary osmidrosis is a common skin disease characterized by an unpleasant odor produced when secretions from apocrine sweat glands in the armpits are decomposed by bacteria on the skin. It affects people's social interactions and psychology. Gold microneedle is a method for treating axillary osmidrosis, which achieves the therapeutic purpose by destroying the glands through radiofrequency heating. However, it remains unknown whether different movement patterns have an impact on the therapeutic effect and adverse reactions.
* Purpose and expected outcomes: This study intends to prospectively collect patients with axillary osmidrosis who visit our hospital, randomly divide them into the horizontal row movement, vertical row movement and mixed movement pattern groups, evaluate the efficacy and occurrence of adverse reactions, and further understand the impact of different microneedle movement patterns on the treatment of axillary osmidrosis.
* Design and methods: Patients who visit our hospital and are willing to receive gold microneedle treatment will be randomly divided into the horizontal row movement, vertical row movement and mixed movement pattern groups. A disposable sterile gold microneedle treatment head will be installed, and different parameters will be set according to the elasticity of the patient's underarm skin and the thickness of subcutaneous fat. The entire radiofrequency treatment area will be covered using horizontal row movement, vertical row movement and mixed movement patterns respectively. All three groups will be closely followed up after the operation; during each follow-up, patients will be required to perform the same exercise load as before the operation to evaluate the therapeutic effect and recurrence.

ELIGIBILITY:
Inclusion criteria: 1) aged from 18 to 50; 2) the axillary odor classified as Grade 2 or 3; 3) without previous history of axillary odor treatment; 4) willingly participated and provided their informed consent.

Exclusion criteria: Patients who met any of the following conditions must be excluded from this study: 1) with other skin diseases in the axilla that may worsen the condition or according to the investigator, may affect the evaluation of the trial results; 2) patients with cicatricial diathesis or needle phobia; 3) patients who were pregnant or lactating; 4) patients with coagulation disorder or immunodeficiency diseases

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2023-10-18 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
cure rate | 6 months

SECONDARY OUTCOMES:
effective rate | 6 months
recurrece rate | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- the First Affiliated Hospital of Chongqing Medical Uiversity, Chongqing, Chongqing Municipality, China